CLINICAL TRIAL: NCT01201317
Title: A Study to Investigate the Analgesic Efficacy of AZD2423 Compared With Placebo
Brief Title: A Study to Investigate the Analgesic Efficacy of AZD2423 Compared With Placebo After 28 Days Treatment in Patients With Painful Diabetic Polyneuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2600C00005
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Neuropathic Pain
Keywords: Analgesic effect
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD2423, 150 mg (Experimental): Tablets, 150 mg once daily in the morning.
  Interventions: Drug: AZD2423
- AZD2423, 20 mg (Experimental): Tablets, 20 mg once daily in the morning.
  Interventions: Drug: AZD2423
- Placebo (Placebo Comparator): Tablets, placebo, once daily in the morning.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2423 — 20 mg tablet
  Arms: AZD2423, 20 mg
Drug: AZD2423 — 150 mg tablet
  Arms: AZD2423, 150 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A study to investigate the analgesic efficacy of AZD2423 compared with placebo after 28 days treatment in patients with painful diabetic polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent form
* Males and female of non-child bearing potential patients aged 18 to 80 years
* Patients with neuropathic pain due to painful diabetic polyneuropathy.

Exclusion Criteria:

* Other pain that may confound assessment of neuropathic pain
* History of treatment failure with more than three adequate trials of medication for neuropathic pain
* Central neuropathic pain conditions (caused by Central Nervous System injury/disease, eg. Stroke)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bror Jonzon, Study Director — AstraZeneca R&D Södertälje
Locations (20):
- United States (14):
  - Research Site, Goodyear, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Los Angeles, California
  - Research Site, DeLand, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sunrise, Florida
  - Research Site, Madisonville, Kentucky
  - Research Site, Willingboro, New Jersey
  - Research Site, New York, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
- Canada (6):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Brampton, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Lachine, Quebec
  - Research Site, Laval

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=204&filename=CSR-D2600C00005.pdf
- See also: CSR-D2600C00005.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=204&filename=CSR-D2600C00005.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on 20th September 2010 and the last participant completed on 6th June 2011. A total of 20 centres in United States (US) and Canada randomised 134 participants.
Pre-assignment Details: The study had an enrolment phase of up to 35 days (including wash-out and baseline periods), a 28-day treatment phase, and a follow-up phase of 7-14 days. Participants were randomly assigned to blinded treatment in a 1:1:1 ratio either to AZD2423 20 mg, AZD2423 150 mg or placebo.
Groups:
- AZD2423 150 mg: tablets, 150 mg once daily in the morning
- AZD2423 20 mg: tablets, 20 mg once daily in the morning
- Placebo: tablets, once daily in the morning
Period: Overall Study
Arm/Group | AZD2423 150 mg | AZD2423 20 mg | Placebo
Started | 48 | 45 | 41
Completed | 39 | 38 | 33
Not Completed | 9 | 7 | 8
Not completed — Withdrawal by Subject | 5 | 0 | 3
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Screen failure | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Study-specific withdrawal criteria | 0 | 0 | 1
Not completed — Painful Diabetic Neuropathy worsening | 0 | 1 | 0
Not completed — Decrease in renal function | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Safety, possible history of tuberculosis | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD2423 150 mg | AZD2423 20 mg | Placebo | Total
Number analyzed (Participants) | 48 | 45 | 41 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (6.9) | 59.6 (8.4) | 56.4 (8.4) | 58 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 20 | 65
  Male | 25 | 23 | 21 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Days 24-28 in Numerical Rating Scale (NRS) Average Pain Score.
Description: Last Observation Carried Forward (LOCF). Twice daily, the participants rated their Average Pain intensity during the past 12 hours on an Numerical Rating Scale (NRS) 0-10; 0=No pain, 10=Worst pain imaginable.
Time Frame: Baseline (mean of Day -5 to Day -1) to the mean of Day 24 to Day 28
Population: Intention-to-treat set (ITT)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD2423 150 mg | AZD2423 20 mg | Placebo
Number analyzed (Participants) | 46 | 42 | 39
Scores on a scale | -1.35 (1.89) | -1.50 (1.77) | -1.61 (2.26)

2. Secondary Outcome: Change From Baseline to Days 24-28 in Numerical Rating Scale (NRS) Worst Pain Score.
Description: Last Observation Carried Forward (LOCF). Twice daily, the participants rated their Worst pain intensity during the past 12 hours on an Numerical Rating Scale (NRS) 0-10, 0=No pain, 10=Worst pain imaginable.
Time Frame: Baseline (mean of Day -5 to Day -1) to the mean of Day 24 to Day 28
Population: Intention-to-treat set (ITT)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD2423 150 mg | AZD2423 20 mg | Placebo
Number analyzed (Participants) | 46 | 42 | 39
Scores on a scale | -1.57 (1.96) | -1.66 (2.06) | -1.80 (2.48)

3. Secondary Outcome: Number of Participants With at Least 30% Decrease From Baseline in Numerical Rating Scale (NRS) Average Pain Score at Day 28.
Description: Last Observation Carried Forward (LOCF). Numerical Rating Scale(NRS) Average Pain score reduction=(change from baseline at Day 28/baseline)*100.
  Responder= NRS Average Pain score reduction ≥30% (yes/no)
Time Frame: Baseline (mean of Day -5 to Day -1) to Day 28
Population: Intention-to-treat set (ITT)
Measure: Number; unit: Participants
Arm/Group | AZD2423 150 mg | AZD2423 20 mg | Placebo
Number analyzed (Participants) | 46 | 42 | 39
Participants | 16 | 19 | 15

4. Secondary Outcome: Number of Participants With at Least 50% Decrease From Baseline in Numerical Rating Scale (NRS) Average Pain Score at Day 28.
Description: Last Observation Carried Forward (LOCF). Numerical Rating Scale (NRS) Average Pain score reduction=(change from baseline at Day 28/baseline)*100.
  Responder= NRS Average Pain score reduction ≥50% (yes/no)
Time Frame: Baseline (mean of Day -5 to Day -1) to Day 28
Population: Intention-to-treat set (ITT)
Measure: Number; unit: Participants
Arm/Group | AZD2423 150 mg | AZD2423 20 mg | Placebo
Number analyzed (Participants) | 46 | 42 | 39
Participants | 10 | 8 | 10

5. Secondary Outcome: Change From Baseline to Day 29 in Neuropathic Pain Symptom Inventory Scale (NPSI) Total Score.
Description: Last Observation carried Forward (LOCF). Scale consists of 10 Neuropathic Pain Symptom Inventory Scale (NPSI) pain symptom descriptors wiht a recall period of 24 hours. Each descriptor is rated on a Numerical Rating Scale (NRS) 0-10; 0=No (symptom), 10=Worst (symptom) imaginable. The NPSI Total Score was calculated as the sum of 10 of the NPSI descriptors. Range for total score 0 -100. Higher total score implicates worse symptoms.
Time Frame: Baseline (Day 1) to Day 29 (Visit 7)
Population: Modified Intention- to- treat set (ITT) including only patients with adequate baseline and Day 29 data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD2423 150 mg | AZD2423 20 mg | Placebo
Number analyzed (Participants) | 35 | 30 | 33
Scores on a scale | -14.63 (22.77) | -12.20 (22.84) | -7.82 (17.02)

ADVERSE EVENTS:
Description: Safety analysis set
Arm/Group | AZD2423 150 mg | AZD2423 20 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/47 | 3/44 | 0/41
Other Adverse Events (participants affected / at risk) | 14/47 | 6/44 | 11/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2423 150 mg (N=47) | AZD2423 20 mg (N=44) | Placebo (N=41)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2423 150 mg (N=47) | AZD2423 20 mg (N=44) | Placebo (N=41)
Headache (Nervous system disorders) | 3 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Pyrexia (General disorders) | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No such publication or presentation may include any of AstraZeneca's Confidential Information without AstraZeneca's prior written approval. AZ should have 60 days for review and can extend time until submission up to 90 days.